CLINICAL TRIAL: NCT02369315
Title: Design of a Multi-site Cluster Randomized Trial to Study the Effects of Musical Training on Child Development in the National System of Child and Youth Orchestras in Venezuela (El Sistema)
Brief Title: Randomized Trial of the Effects of Musical Training on Child Development in the Venezuela Orchestra Program (El Sistema)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inter-American Development Bank (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: IDB-2014-VE-1
Record Dates: First submitted 2015-02-16; First posted 2015-02-23 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Child Development
Keywords: child development; music training; self-regulation; exposure to violence
MeSH Terms: conditions — Self-Control | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Invited entry 2012) (Experimental): Children offered entry to music program in September 2012
  Interventions: Behavioral: Treatment (Invited entry 2012)
- Control (Invited entry 2013) (Experimental): Children offered entry to music program delayed until September 2013
  Interventions: Behavioral: Control (Invited entry 2013)

INTERVENTIONS:
Behavioral: Treatment (Invited entry 2012) — Entry to music program offered in September 2012
  Arms: Treatment (Invited entry 2012)
Behavioral: Control (Invited entry 2013) — Entry to music program offered in September 2013
  Arms: Control (Invited entry 2013)

SUMMARY:
This study evaluates Venezuela's National System of Child and Youth Orchestras, better known as "El Sistema".

DETAILED DESCRIPTION:
The randomized control trial was conducted in 16 music centers in Venezuela between May 2012 and November 2013, with a population of 6-14 year olds seeking entry to the program. During an application period (May-July 2012), 2,603 guardians (the experimental cluster) applied on behalf of 2,999 6-14 year olds. Approximately half of the guardians were randomly offered early admission in September 2012, with the rest offered admission in September 2013. Baseline and follow-up data were collected on outcomes which will be explored for full-group and specific sub-groups (children with less educated mothers, and boys or girls exposed to violence).

ELIGIBILITY:
Inclusion criteria:

* Excess demand in 5 geographic areas: 24 music centers across the 5 states were identified as the experimental sites based on the likelihood of having excess demand by families in the 2012-13 academic year.
* Apply protocol: Experimental sites agreed to accept written applications from guardians between May 7 and July 8, 2012 (without informing guardians of admission decisions until after randomization). Directors consented to participate in the experiment and received training in the experimental protocol. Children were eligible to apply if they would be 6 to 14 years old on September 1, 2012. Sites received applications from 2,603 guardians on behalf of 2,999 children.

Exclusion criteria:

* Music center level: Two sites were excluded because their directors declined to follow the experimental protocol, and six were excluded because of insufficient demand to carry out randomized experiment.
* Child/guardian level: By prior agreement, each site director could award early admission to a small number of applicants (no more than 5% of positions). In eight sites, 85 children (of 74 guardians) were excluded from the study because they entered through these positions allotted to site directors. Children were also lost from study if parental consent and child assent not given.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2914 (Actual)
Dates: Start 2012-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Child self-regulatory skills | 1 year (baseline 2012 to followup 2013)
  self-reported 10 item self-control scale; response inhibition (Go/no-go), attention functioning (Flanker), and planning skills (Tower of London)
Child Behaviors | 1 year (baseline 2012-followup 2013)
  prosocial behavior (SDQ Strengths subscale), difficulties (SDQ Difficulties subscale), risk-taking (risky driving game), and aggression (aggressive behavior and propensity scales)
Child Prosocial Skills and Connections | 1 year
  child self-esteem (Rosenberg scale), empathy (Bryant scale), and school and family engagement (BERS-2 subscales)
Child Cognitive Skills | 1 year (baseline 2012-followup 2013)
  working memory (digit recall), processing speed (symbol search), and visual-spatial reasoning (Raven)

SECONDARY OUTCOMES:
Guardian Collective Efficacy | 1 year (baseline 2012-followup 2013)
  collective efficacy scale of Sampson et. al. 1997

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Duryea, Ph.D., Principal Investigator — Inter-American Development Bank; Patrick McEwan, Ph.D., Principal Investigator — Wellesley College; Nancy Guerra, Ph.D., Principal Investigator — University of Delaware; Marco Stampini, Ph.D., Principal Investigator — Inter-American Development Bank

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aleman X, Duryea S, Guerra NG, McEwan PJ, Munoz R, Stampini M, Williamson AA. The Effects of Musical Training on Child Development: a Randomized Trial of El Sistema in Venezuela. Prev Sci. 2017 Oct;18(7):865-878. doi: 10.1007/s11121-016-0727-3. PMID 27896644
- See also: The Effects of Musical Training on Child Development: a Randomized Trial of El Sistema in Venezuela — http://rd.springer.com/article/10.1007/s11121-016-0727-3